CLINICAL TRIAL: NCT02997865
Title: Stepped Care for Depression in Heart Failure
Acronym: DASH-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01HL131524 (NIH); R01HL131524 (NIH)
Record Dates: First submitted 2016-12-15; First posted 2016-12-20 (Estimated); Results first posted 2023-02-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-01

CONDITIONS: Heart Failure; Depressive Disorder, Major
Keywords: heart failure; depressive disorder, major; cognitive therapy; self-care
MeSH Terms: conditions — Heart Failure; Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stepped Care for Depression (Experimental): Participants will receive cognitive behavior therapy for depression, plus referral to their own physician for discussion of antidepressant medication if symptoms do not improve within 5-10 weeks. Participants will also receive individually-tailored heart failure self-care education and support.
  Interventions: Behavioral: Stepped care for depression
- Enhanced Usual Care (No Intervention): Participants will receive individually-tailored heart failure self-care education and support. With the participant's permission, his or her personal physician will be notified about the patient's depression. The participant will be asked to discuss depression treatment options with his or her personal physician.

INTERVENTIONS:
Behavioral: Stepped care for depression — Cognitive behavior therapy (CBT), plus referral to the participant's own physician to discuss antidepressant medications if indicated.
  Arms: Stepped Care for Depression

SUMMARY:
This study evaluates stepped care for depression in patients with heart failure (HF). The stepped care intervention consists of individualized cognitive behavior therapy (CBT). Half of the participants will receive stepped care and half will receive usual care for depression; all participants will receive heart failure self-care education and support. The primary aims are to determine whether stepped care is superior to usual care for depression, and whether treating depression improves heart failure self-care outcomes.

DETAILED DESCRIPTION:
Depression is associated with poor heart failure self-care. Good self-care practices, including following dietary recommendations, taking prescribed medications, monitoring symptoms, and regular light exercise have been shown to improve quality of life and survival in persons with heart failure.

Both CBT and antidepressant medications have been used in previous studies to treat major depression in patients with heart failure. Participants in the intervention arm in this trial will start with CBT. Those who do not improve very much within the first 5-10 weeks of CBT may also be referred to their own physician to discuss antidepressant medications.

Heart failure self-care education and support will be provided after the first 8 weeks of the depression intervention. The study will determine whether people with heart failure benefit more from self-care education and support after their depression has been treated with a stepped care intervention, as compared to usual care for depression as provided by primary care providers.

ELIGIBILITY:
Inclusion Criteria:

1. Stable, clinically-documented New York Heart Association (NYHA) Class I-III heart failure.
2. Current major depressive episode.
3. Baseline Beck Depression Inventory (BDI-II) score 14 or greater

Exclusion Criteria:

1. Dementia or other significant cognitive or communication deficits
2. Terminal illness other than HF
3. Insurmountable logistical barriers to participation
4. Age less than 25 years
5. Current clinically significant substance abuse, bipolar disorder, schizophrenia, or other psychotic disorder
6. High risk of suicide
7. Current participation in non-study psychotherapy for depression or other psychiatric conditions
8. Initiation or modification of antidepressant medication treatment within past two months
9. Renal or hepatic conditions that would preclude the use of antidepressants.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2017-02-17 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth E Freedland, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Behavioral Medicine Center Washington University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
We may share de-identified data with other researchers after the completion of the study; no specific plans for this have been made yet.
Supporting Information: Study Protocol, SAP
Time Frame: Mid-2022 through 2023
Access Criteria: Permission of Principal Investigator

REFERENCES:
- [Result] Freedland KE, Skala JA, Carney RM, Steinmeyer BC, Rubin EH, Rich MW. Sequential Interventions for Major Depression and Heart Failure Self-Care: A Randomized Clinical Trial. Circ Heart Fail. 2022 Aug;15(8):e009422. doi: 10.1161/CIRCHEARTFAILURE.121.009422. Epub 2022 Jun 21. PMID 35973032
- [Derived] Freedland KE, Skala JA, Carney RM, Steinmeyer BC, Rich MW. Outcomes of a tailored self-care intervention for patients with heart failure and major depression: A secondary analysis of a randomized controlled trial. Int J Nurs Stud. 2023 Nov;147:104585. doi: 10.1016/j.ijnurstu.2023.104585. Epub 2023 Aug 9. PMID 37611354
- [Derived] Freedland KE, Skala JA, Carney RM, Steinmeyer BC, Rich MW. Treatment of depression and inadequate self-care in patients with heart failure: One-year outcomes of a randomized controlled trial. Gen Hosp Psychiatry. 2023 Sep-Oct;84:82-88. doi: 10.1016/j.genhosppsych.2023.06.001. Epub 2023 Jun 7. PMID 37406374

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between February 2017 and January 2021, patients who had a clinical diagnosis of NYHA Class I-III heart failure and who received medical care at Washington University Medical Center in St. Louis were screened for study eligibility. Those who were younger than 25 years of age or who were too ill or cognitively impaired to participate were excluded. Eligible patients who provided written informed consent were enrolled.
Groups:
- Stepped Care for Depression: Participants will receive cognitive behavior therapy for depression, plus referral to their own physician for discussion of antidepressant medication if symptoms do not improve within 5-10 weeks. Participants will also receive individually-tailored heart failure self-care education and support, i.e., a Tailored Self-Care (TSC) intervention.
  Stepped care for depression: Cognitive behavior therapy (CBT), plus referral to the participant's own physician to discuss antidepressant medications if indicated.
- Enhanced Usual Care: Participants will receive individually-tailored heart failure self-care education and support, i.e., a Tailored Self-Care (TSC) intervention. With the participant's permission, his or her personal physician will be notified about the patient's depression. The participant will be asked to discuss depression treatment options with his or her personal physician.
Period: Overall Study
Arm/Group | Stepped Care for Depression | Enhanced Usual Care
Started | 69 | 70
Completed | 56 (Number of participants who completed the Week 32 outcome assessments.) | 66 (Number of participants who completed the Week 32 outcome assessments.)
Not Completed | 13 | 4
Not completed — Death | 2 | 1
Not completed — Lost to Follow-up | 6 | 3
Not completed — Withdrawal by Subject | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stepped Care for Depression | Enhanced Usual Care | Total
Number analyzed (Participants) | 69 | 70 | 139
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.0 (11.5) | 58.3 (12.2) | 58.2 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 35 | 68
  Male | 36 | 35 | 71
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 67 | 69 | 136
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 34 | 29 | 63
  White | 34 | 32 | 66
  More than one race | 1 | 7 | 8
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 69 | 70 | 139
Education (12 years or less) [Count of Participants; unit: Participants] | 17 | 14 | 31
Income ($30,000/year or less) [Count of Participants; unit: Participants] | 35 | 30 | 65
Married or partnered [Count of Participants; unit: Participants] | 26 | 27 | 53
Left ventricular ejection fraction <45% [Count of Participants; unit: Participants] | 36 | 41 | 77
New York Heart Association (NYHA) class [Count of Participants; unit: Participants] — NYHA class indicates the functional or symptomatic severity of heart failure. Class I indicates asymptomatic (i.e., best class), class IV indicates severe heart failure (patient is unable to engage in normal physical activities), and classes II and II represent intermediate levels of functional impairment or symptom severity. Lower NYHA ratings represent better functioning or milder symptoms. Participants were classified at baseline as NYHA class I-II vs. class III-IV. The table values refer to the number and column percentage of patients in class I-II.
  Participants | 44 | 47 | 91
Antidepressant medication [Count of Participants; unit: Participants] | 31 | 31 | 62
Patient Health Questionnaire (PHQ-9) [Mean (Standard Deviation); unit: units on a scale] — The Patient Health Questionnaire (PHQ-9) is a 9-item patient self-report questionnaire that assesses the presence and severity of major depression. Each item represents one of the Diagnostic and Statistical Manual (DSM-5) symptoms of major depression. The item ratings range in symptom frequency from 0 (absent) to 3 (nearly every day). Scores of 5, 10, 15, and 20 represent cutpoints for mild, moderate, moderately severe and severe depression, respectively. Total scores on the PHQ-9 can range from 0 to 27. Lower PHQ-9 scores represent better outcomes.
  units on a scale | 16.9 (4.7) | 16.2 (5.3) | 16.5 (5.0)
Beck Depression Inventory (BDI-2) [Mean (Standard Deviation); unit: units on a scale] — The Beck Depression Inventory (BDI-2) is a 21-item patient self-report measure of the severity of depression. Each item is rated on a 4-point scale ranging from 0 to 3. The minimum total score is zero and the maximum total score is 63. A total score of 0-13 is considered nondepressed, 14-19 represents mild depression, 20-28 represents moderate depression, and 29-63 represents severe depression. Lower scores represent better outcomes.
  units on a scale | 32.6 (8.3) | 32.1 (9.2) | 32.3 (8.8)
Hamilton Rating Scale for Depression (HAM-D-17) [Mean (Standard Deviation); unit: units on a scale] — The Hamilton Rating Scale for Depression (HAM-D-17) is a 17-item interviewer-rated measure of the severity of depression. The total score is created by summing the item ratings. Total scores can range from zero to 52. Scores of 0-7 are considered to be in the nondepressed range, 8-16 indicate mild depression, 17-23 indicate moderate depression, and scores over 24 indicate severe depression. Lower scores represent better outcomes.
  units on a scale | 22.5 (5.6) | 22.6 (5.4) | 22.6 (5.5)
Self-Care of Heart Failure Index: Maintenance [Mean (Standard Deviation); unit: units on a scale] — The 10-item Self-Care of Heart Failure (SCHFI v6.2) Maintenance scale assesses the frequency of engagement in heart failure-related health behaviors. The total score is standardized and can range from 0 (worst) to 100 (best). Adequate self-care maintenance behavior is defined as a score of 70 or higher
  units on a scale | 60.7 (15.7) | 55.5 (16.2) | 58.1 (16.1)
Self-Care of Heart Failure Index: Management [Mean (Standard Deviation); unit: units on a scale] — The 6-item Self-Care of Heart Failure (SCHFI v6.2) Management scale assesses the patient's responses to signs or symptoms of acute or worsening heart failure. The total score is standardized and can range from 0 (worst) to 100 (best). Adequate self-care management behavior is defined as a score of 70 or higher.
  units on a scale | 55.7 (22.2) | 52.4 (22.6) | 52.4 (22.0)
Self-Care of Heart Failure Index: Confidence [Mean (Standard Deviation); unit: units on a scale] — The 6-item Self-Care of Heart Failure (SCHFI v6.2) Confidence scale assesses the patient's confidence in his/her ability to manage the signs and symptoms of heart failure. The total score is standardized and can range from 0 (worst) to 100 (best). Adequate self-care confidence behavior is defined as a score of 70 or higher.
  units on a scale | 58.8 (23.7) | 51.0 (23.3) | 54.8 (23.7)
Beck Anxiety Inventory (BAI) [Mean (Standard Deviation); unit: units on a scale] — The Beck Anxiety Inventory (BAI) is a 21-item patient-self report questionnaire about symptoms of anxiety. Each symptom is rated on a four-point scale ranging from 0 (not at all) to 3 (severe - it bothered me a lot). Total scores can range from 0 (best) to 63 (worst). Scores of 0-21 indicate little or no anxiety, 22-35 moderate anxiety, and 36-63 severe anxiety.
  units on a scale | 23.2 (12.3) | 22.1 (13.2) | 22.7 (12.7)
Kansas City Cardiomyopathy Questionnaire (KCCQ) [Mean (Standard Deviation); unit: units on a scale] — The 12-item Kansas City Cardiomyopathy Questionnaire (KCCQ) overall summary score is scaled to range from 0 (worst) to 100 (best) heart-failure-related quality of life. Scores of 0 to 24 represent very poor to poor qualify to life; 25 to 49 poor to fair quality of life; 50 to 74 fair to good quality of life; and 75 to 100 good to excellent quality of life.
  units on a scale | 45.9 (22.0) | 46.5 (18.9) | 46.2 (20.4)

OUTCOME MEASURES:

1. Primary Outcome: Beck Depression Inventory (BDI-2) Total Score
Description: The BDI-2 was used to assess the patient's self-reported severity of depression. Total scores can range from zero (best) to 63 (worst). Scores between 0-13 are considered to be in the nondepressed range; 14-19 are consistent with mild, 20-28 with moderate, and 29-63 with severe depression.
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stepped Care for Depression | Enhanced Usual Care
Number analyzed (Participants) | 69 | 70
score on a scale | 15.6 (9.7) | 19.6 (9.4)

2. Primary Outcome: Self Care of Heart Failure Index (SCHFI) Maintenance Subscale
Description: The SCHFI Maintenance scale assesses self-reported heart failure self-care behaviors. The Maintenance score was the trial's primary self-care outcome measure. Scores range from 0 (worst) to 100 (best), with scores of 70 or higher consistent with adequate self-care.
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stepped Care for Depression | Enhanced Usual Care
Number analyzed (Participants) | 69 | 70
score on a scale | 70.4 (12.5) | 73.0 (11.6)

3. Secondary Outcome: Beck Anxiety Inventory
Description: The BAI measures the self-reported severity of anxiety symptoms. Total BAI scores range from 0 (best) to 63 (worst). A total score of 0-7 is considered nonanxious; scores between 8-15 are consistent with mild, 16-25 moderate, and 26-63 severe anxiety.
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stepped Care for Depression | Enhanced Usual Care
Number analyzed (Participants) | 69 | 70
score on a scale | 12.5 (9.3) | 15.1 (8.9)

4. Secondary Outcome: Kansas City Cardiomyopathy Questionnaire (KCCQ)
Description: The KCCQ assesses the patient's self-reported, heart failure-related functioning and quality of life. Scores range from 0 (worst) to 100 (best). Scores between 0-24 are consistent with very poor to poor health status, 25-49 poor to fair health status, 50-74 fair to good health status, and 75-100 good to excellent health status.
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stepped Care for Depression | Enhanced Usual Care
Number analyzed (Participants) | 69 | 70
score on a scale | 63.7 (16.9) | 61.2 (57.0)

5. Secondary Outcome: Hamilton Rating Scale for Depression (HAM-D-17)
Description: The Hamilton Rating Scale total score indicates the interviewer-rated severity of depression symptoms. Total scores can range from 0 to 52, with higher scores indicating worse depression. Patients who score 0-9 are considered to be nondepressed. Scores of 10-13 represent mild, 14-17 mild to moderate, and >17 moderate to severe depression.
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stepped Care for Depression | Enhanced Usual Care
Number analyzed (Participants) | 69 | 70
score on a scale | 12.5 (5.7) | 15.0 (4.9)

6. Secondary Outcome: Actigraphy
Description: Actigraphy was used to track the patient's physical activity level. However, actigraphy had to be discontinued during the first few months of the trial due to the COVID-19 pandemic.
Time Frame: 16 weeks
Population: Although we planned to collect actigraphy data at baseline and 16 weeks and report the 16-week data as an outcome, we were unable to collect actigraphy data due to the coronavirus (COVID-19) pandemic.
Arm/Group | Stepped Care for Depression | Enhanced Usual Care
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 32 weeks
Description: All-cause mortality. Obtained from hospitalization records, informant interviews, online records, or other sources.
Arm/Group | Stepped Care for Depression | Enhanced Usual Care
All-Cause Mortality (participants affected / at risk) | 4/69 | 1/70
Serious Adverse Events (participants affected / at risk) | 0/69 | 0/70
Other Adverse Events (participants affected / at risk) | 0/69 | 0/70

LIMITATIONS AND CAVEATS:
This was a single-center trial. Fewer patients were enrolled than planned, primarily due to recruitment challenges during the COVID-19 pandemic. Actigraphy data could not be collected due to the pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-08-26): https://cdn.clinicaltrials.gov/large-docs/65/NCT02997865/Prot_001.pdf
  • Statistical Analysis Plan (2021-08-24): https://cdn.clinicaltrials.gov/large-docs/65/NCT02997865/SAP_002.pdf